CLINICAL TRIAL: NCT03238417
Title: Evaluating Evidence-Based Quality Improvement of Comprehensive Women's Health Care Implementation in Low-Performing VA Facilities (PEC 16-352)
Brief Title: Evaluating Evidence-Based Quality Improvement of Comprehensive Women's Health Care Implementation in Low-Performing VAs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: PEX 16-002; PEC 16-352 (Other Grant/Funding Number: QUERI Program)
Record Dates: First submitted 2017-07-25; First posted 2017-08-03 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Comprehensive Care
Keywords: women's health; primary health care; mental health; Veterans; quality improvement
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Dynamic waitlist control design with a group of 7 VA facilities was randomly allocated to Evidence-Based Quality Improvement (EBQI) in Year 1 (while 14 VA facilities serving as waitlist controls), the second group of 7 VA facilities was randomly allocated to EBQI in Year 2 (while the 7 remaining VA facilities and the first 7 EBQI sites serving as control), and the final group of 7 VA facilities was randomly allocated to EBQI in Year 3 (while the first 14 EBQI facilities subsequently serving as control). By the end of the three year study period, a total of 21 VA facilities received at least 1 year of EBQI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evidence-Based Quality Improvement (EBQI) (Experimental): EBQI represents a multilevel stakeholder engaged top-down/bottom-up research-clinical partnership approach to systematically improving the design and implementation of local innovations adapted to local contexts. The EBQI contractor will (1) convene facility-level stakeholder meetings, (2) facilitate local facility-level QI team design meetings, (3) provide external practice facilitation through within and across facility QI collaboration calls, (4) provide formative QI data feedback and (5) provide QI training/education to local teams.
  Interventions: Other: Evidence-Based Quality Improvement
- Waitlist Controls (No Intervention): Waitlist controls will continue naturalistic routine care implementation of VHA directives and other guidance related to comprehensive women's health care.

INTERVENTIONS:
Other: Evidence-Based Quality Improvement — Multilevel research-clinical partnership approach to supporting local strategic planning, priority setting, skill building and engagement in addressing targeted healthcare delivery problems. Launched at participating VA facilities through advance key stakeholder interviews, in-person site visits, data review (e.g., structure and environment of care, gender disparities in quality and patient experience), QI education/training, technical support (e.g., QI project and measures development), additional formative feedback from the evaluation (e.g., provider/survey measure summaries), external and internal practice facilitation, and across-EBQI site collaboration calls. Local leadership, EBQI champions and QI teams develop and implement innovation projects aimed at improving prioritized quality targets related to women Veterans' health and healthcare needs as well as facility-level structural changes needed to improve compliance with VA guidelines.
  Other Names: EBQI
  Arms: Evidence-Based Quality Improvement (EBQI)

SUMMARY:
Gaps in delivery of gender-sensitive comprehensive care have resulted in disparities in quality and patient experience among women seen in VA. VA policy action providing guidance on delivery of comprehensive healthcare services for women Veterans was disseminated nationally in 2010, followed by annual assessments and site visits evaluating local VA efforts. While substantial inroads have been made, policy implementation, even when leveraged by field-based women's health leaders, has not been uniformly successful in achieving delivery of comprehensive care by designated providers in gender-sensitive care environments that ensure women's privacy, dignity and safety, all tenets of the original guidance and the updated directive (2017).

Building on prior effectiveness of an evidence-based quality improvement (EBQI) approach to tailoring VA's medical home model -- Patient Aligned Care Teams (PACT) -- to the needs of women Veterans, VA leaders in women's health adopted EBQI to help low-performing VAs systematically improve services.

The objectives of the resulting Partnered Evaluation Initiative (PEI) funded by VA's Quality Enhancement Research Initiative and VA Office of Women's Health were:

1. To evaluate barriers and facilitators to achieving delivery of comprehensive women's health care in the identified low-performing VAs;
2. To evaluate effectiveness of EBQI in supporting low-performing VA facilities achieve improved organizational features, provider/staff attitudes, quality of care, and patient experiences among women Veteran patients; and,
3. To evaluate contextual factors, local implementation processes, and organizational changes in the participating facilities over time.

DETAILED DESCRIPTION:
Gaps in delivery of gender-sensitive comprehensive care have resulted in disparities in quality and patient experience among women seen in VA. VA policy action providing guidance on delivery of comprehensive healthcare services for women Veterans was disseminated nationally in 2010, followed by annual assessments and site visits evaluating local VA efforts. While substantial inroads have been made, policy implementation, even when leveraged by field-based women's health leaders, has not been uniformly successful in achieving delivery of comprehensive care by designated providers in gender-sensitive care environments that ensure women's privacy, dignity and safety, all tenets of the original guidance and the updated VA directive (2017).

In collaboration with VA Women's Health Services (WHS), VA researchers developed a series of studies to better understand and help improve comprehensive care implementation through the Women Veterans' Healthcare CREATE Initiative. Among these, one focused on testing an evidence-based quality improvement (EBQI) approach to tailoring VA's medical home model -- Patient Aligned Care Teams (PACT) -- to the needs of women Veterans, which has yielded significant local improvements in women Veterans' care. EBQI emphasizes a multilevel partnered approach to building capacity for innovation, implementation and spread of evidence-based practice. With its demonstrated success in the CREATE PACT study and several other EBQI trials, WHS adopted EBQI as a strategy to help low-performing VA facilities systematically improve services.

The objectives of the WHS/QUERI Partnered Evaluation Initiative that this project represents are:

1. To evaluate the barriers and facilitators to achieving delivery of comprehensive women's health care in the identified low-performing VA facilities;
2. To evaluate the effectiveness of EBQI in supporting low-performing VA facilities achieve improved:

   1. Organizational features (e.g., level of comprehensive services available; care coordination arrangements; PACT features implemented; environment of care improvements);
   2. Provider/staff attitudes (e.g., improved gender awareness; women's health knowledge and practice);

   d) Quality of care and patient experiences among women Veteran patients using secondary data; and,
3. To evaluate contextual factors, local implementation processes, and organizational changes in the participating facilities over time.

Results of the evaluation have been used to provide feedback to stakeholders, including women Veterans, at the local, network and national levels, while also being used to continuously refine EBQI implementation processes. The evaluation is also helping inform optimal strategies for ongoing improvements in women Veterans' care in the 21 participating VA facilities, other VA facilities and for other improvement initiatives in this and other national program offices.

ELIGIBILITY:
Inclusion Criteria:

* Unit of randomization: VA healthcare facilities (VA medical center or community-based outpatient clinic)
* Subset of VA healthcare facilities identified as low-performing on the basis of composites of access/wait times, gender disparities in quality, e.g.:

  * depression screening
  * diabetic blood sugar control
* Presence/absence of VA-required structural facets of care, e.g.:

  * designated women's health providers
  * mammography coordinator
  * gynecology access
  * Women Veteran Program Manager (WVPM)
  * 3:1 staffing ratio for PACT teamlets

Key Stakeholder Inclusion Criteria (qualitative interviews):

* Veteran Integrated Service Network (VISN) level leader (Director or Chief Medical Officer)
* VISN level WVPM Lead, VISN level primary care director, VISN level QI/system redesign lead)
* VA facility leader (Director or other member of senior leadership)
* Chief of Staff
* primary care director
* women's health medical director
* WVPM
* local EBQI champion
* other key personnel

Provider/Staff Survey Inclusion Criteria:

* Primary care providers (medical doctor [MD], doctor of osteopathy [DO], nurse practitioner [NP], physician assistant [PA]) delivering primary care in general primary care and/or women's health clinics
* PACT teamlet members (registered nurse [RN] care managers, licensed vocational nurse/licensed practical nurse [LVN/LPN]/health technicians, and clerks)
* larger PACT team members, e.g.:

  * social workers
  * dieticians
  * health coaches
  * integrated mental health

Exclusion Criteria:

* Facility-level exclusion: Facilities not identified in the initial sample of VA facilities (sample not renewed over time).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Yano, PhD MSPH, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA; Alison B Hamilton, PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (25):
- United States (25):
  - Central Alabama Veterans Health Care System West Campus, Montgomery, AL, Montgomery, Alabama
  - Northern Arizona VA Health Care System, Prescott, AZ, Prescott, Arizona
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Carl Vinson VA Medical Center, Dublin, GA, Dublin, Georgia
  - Marion VA Medical Center, Marion, IL, Marion, Illinois
  - Robert J. Dole Department of Veterans Affairs Medical and Regional Office Center, Wichita, KS, Wichita, Kansas
  - Overton Brooks VA Medical Center, Shreveport, LA, Shreveport, Louisiana
  - Rehabilitation R&D Service, Baltimore, MD, Baltimore, Maryland
  - Battle Creek VA Medical Center, Battle Creek, MI, Battle Creek, Michigan
  - Harry S. Truman Memorial, Columbia, MO, Columbia, Missouri
  - VA Southern Nevada Healthcare System, North Las Vegas, NV, Las Vegas, Nevada
  - Bath VA Medical Center, Bath, NY, Bath, New York
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Chalmers P. Wylie Ambulatory Care Center, Columbus, OH, Columbus, Ohio
  - VA Black Hills Health Care System Fort Meade Campus, Fort Meade, SD, Fort Meade, South Dakota
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas
  - Hampton VA Medical Center, Hampton, VA, Hampton, Virginia
  - Jonathan M. Wainwright Memorial VA Medical Center, Walla Walla, WA, Walla Walla, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamilton AB, Olmos-Ochoa TT, Canelo I, Rose D, Hoggatt KJ, Than C, Yano EM. Dynamic waitlisted design for evaluating a randomized trial of evidence-based quality improvement of comprehensive women's health care implementation in low-performing VA facilities. Implement Sci Commun. 2020 Jun 30;1:59. doi: 10.1186/s43058-020-00038-0. eCollection 2020. PMID 32885214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cross-sectional surveys were sent to primary care providers and staff at 21 VA Medical Centers at baseline, 12 months, and 24 months.
Pre-assignment Details: Twenty one VA facilities were randomized to receive evidence-based quality improvement (EBQI) in a dynamic waitlist control design in which seven facilities received EBQI per year while the remaining 14 facilities were assigned as control.
Units Other Than Participants: VA Medical Centers
Groups:
- Evidence-Based Quality Improvement (EBQI): EBQI represents a multilevel stakeholder engaged top-down/bottom-up research-clinical partnership approach to systematically improving the design and implementation of local innovations adapted to local contexts. The EBQI contractor will (1) convene facility-level stakeholder meetings, (2) facilitate local facility-level quality improvement (QI) team design meetings, (3) provide external practice facilitation through within and across facility QI collaboration calls, (4) provide formative QI data feedback and (5) provide QI training/education to local teams.
  Launched at participating VA facilities through advance key stakeholder interviews, in-person site visits, data review (e.g., structure and environment of care, gender disparities in quality and patient experience), QI training, technical support (e.g., QI project and measures development), additional formative feedback from the evaluation (e.g., provider/survey measure summaries), external and internal practice facilitation, and across-EBQI site collaboration calls. Local leadership, EBQI champions and QI teams develop and implement innovation projects aimed at improving prioritized quality targets related to women Veterans' health and healthcare needs as well as facility-level structural changes needed to improve compliance with VA guidelines.
- Waitlist Controls: Waitlist controls will continue naturalistic routine care implementation of VA directives and other guidance related to comprehensive women's health care.
Period: Overall
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Started | 1330; 7 VA Medical Centers | 2632; 14 VA Medical Centers
Completed | 327; 7 VA Medical Centers | 644; 14 VA Medical Centers
Not Completed | 1003; 0 VA Medical Centers | 1988; 0 VA Medical Centers
Not completed — non-response | 955 | 1920
Not completed — partial completion | 48 | 68
Period: Baseline
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Started | 513; 7 VA Medical Centers | 934; 14 VA Medical Centers
Completed | 124; 7 VA Medical Centers | 217; 14 VA Medical Centers
Not Completed | 389; 0 VA Medical Centers | 717; 0 VA Medical Centers
Not completed — Partial completion | 17 | 48
Not completed — non-response | 372 | 669
Period: 12-month
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Started | 400; 7 VA Medical Centers | 911; 14 VA Medical Centers
Completed | 81; 7 VA Medical Centers | 205; 14 VA Medical Centers
Not Completed | 319; 0 VA Medical Centers | 706; 0 VA Medical Centers
Not completed — non-response | 296 | 669
Not completed — partial completion | 23 | 37
Period: 24-month
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Started | 417; 7 VA Medical Centers | 847; 14 VA Medical Centers
Completed | 122; 7 VA Medical Centers | 222; 14 VA Medical Centers
Not Completed | 295; 0 VA Medical Centers | 625; 0 VA Medical Centers
Not completed — non-response | 287 | 594
Not completed — partial completion | 8 | 31

BASELINE CHARACTERISTICS:
Population: primary care providers and staff
Units Other Than Participants: VA Medical Centers
Groups:
- Evidence-Based Quality Improvement (EBQI): EBQI represents a multilevel stakeholder engaged top-down/bottom-up research-clinical partnership approach to systematically improving the design and implementation of local innovations adapted to local contexts. The EBQI contractor will (1) convene facility-level stakeholder meetings, (2) facilitate local facility-level QI team design meetings, (3) provide external practice facilitation through within and across facility QI collaboration calls, (4) provide formative QI data feedback and (5) provide QI training/education to local teams.
  Launched at participating VA facilities through advance key stakeholder interviews, in-person site visits, data review (e.g., structure and environment of care, gender disparities in quality and patient experience), QI training, technical support (e.g., QI project and measures development), additional formative feedback from the evaluation (e.g., provider/survey measure summaries), external and internal practice facilitation, and across-EBQI site collaboration calls. Local leadership, EBQI champions and QI teams develop and implement innovation projects aimed at improving prioritized quality targets related to women Veterans' health and healthcare needs as well as facility-level structural changes needed to improve compliance with VA guidelines.
- Total: Total of all reporting groups
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls | Total
Number analyzed (Participants) | 124 | 217 | 341
Number analyzed (VA Medical Centers) | 7 | 14 | 21
Age, Customized [Count of Participants; unit: Participants]
  age: 20-29 | 1 | 8 | 9
  age: 30-39 | 16 | 39 | 55
  age: 40-49 | 23 | 53 | 76
  age: 50-59 | 51 | 64 | 115
  age: 60+ | 16 | 26 | 42
  age: missing | 17 | 27 | 44
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 91 | 163 | 254
  Gender: Male | 17 | 30 | 47
  Gender: missing | 16 | 24 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Primary care provider and staff [Count of Participants; unit: Participants]
  Primary care providers | 23 | 50 | 73
  staff | 101 | 167 | 268
Years worked in VA [Mean (Standard Deviation); unit: years] | 9.85 (8.40) | 6.96 (7.24) | 8.01 (7.79)

OUTCOME MEASURES:

1. Primary Outcome: Gender-sensitive Care Environment
Description: Multi-item scale score reflecting survey items (from The Women's Assessment Tool for Comprehensive Health (WATCH)) on availability of same-gender providers, availability of same-gender staff, privacy of physical layout, availability of privacy curtains, level of implementation of local culture campaign that values and treats Women Veterans with respect. The score ranges from 0 to 7, with a higher score reflecting greater gender-sensitive care environment.
Time Frame: 12-month change in gender-sensitive care environment
Population: One Women Veteran Program Manger per VA Medical Center responded to the survey about the site's Women's Health Program on WATCH.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: VA Medical Centers.
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 7 | 14
Number analyzed (VA Medical Centers.) | 7 | 14
score on a scale
  Baseline | 4.2 (2.3) | 3.3 (1.9)
  12 month | 1.6 (1.9) | 1.4 (1.7)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — Analysis of Variance comparing change in outcome between EBQI and control from baseline to 12 month; p = 0.623, ANOVA — P-value is from the interaction term between EBQI and time; Mean Difference (Net) = -0.65, 95% CI 2-sided [-3.3 to 2.0], Standard Error of Mean 1.32

2. Primary Outcome: Gender-sensitive Care Environment
Description: as for outcome 1
Time Frame: 24-month change in gender-sensitive care environment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: VA Medical Center
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 7 | 14
Number analyzed (VA Medical Center) | 7 | 14
score on a scale
  Baseline | 4.2 (2.3) | 3.3 (1.9)
  24 month | 3.2 (0.8) | 2.8 (1.6)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — Analysis of Variance testing for change in outcome between EBQI and control from baseline to 24 months; p = 0.678, ANOVA — P-value is from the interaction term of EBQI and time; Mean Difference (Net) = -0.48, 95% CI 2-sided [-2.8 to 1.8], Standard Error of Mean 1.1

3. Primary Outcome: Gender Awareness
Description: A 12-item score reflecting primary care and women's health providers' and staff's awareness and knowledge of women Veterans' military background and healthcare needs. The score ranges from 1 to 5 with higher scores reflecting greater gender awareness.
Time Frame: 12-month change in gender awareness among VA primary care and women's health providers and staff.
Population: Primary care and women's health providers and staff. The analysis was based on cases with non-missing outcome data. There are 19 missing cases in the EBQI arm and 39 missing in the control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 205 | 422
Number analyzed (VA Medical Centers) | 7 | 14
score on a scale
  baseline | 3.66 (0.53) | 3.63 (0.49)
  12- month | 3.67 (0.61) | 3.62 (0.52)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Change in gender awareness score between EBQI and control from baseline to 12-month; Test type: Superiority — Difference-in-differences analysis using linear regression, adjusted for age, how often they saw women patients in the past year, location of practice in primary care or women's health clinic, and having had any type of quality improvement training. We adjusted our analysis with non-response weights; p = 0.364, Regression, Linear — P-value is from the interaction term between EBQI and time, adjusted for non-response weights and characteristics described in the statistical analysis overview; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.17 to 0.35], Standard Error of Mean 0.13 — The estimated value reported here is the predicted mean change from baseline to 12-month, adjusting for characteristics described in the statistical analysis overview

4. Primary Outcome: Gender Awareness
Description: A 12-item score reflecting primary care and women's health providers' and staff's awareness and knowledge of women Veterans' military roles and healthcare needs . The score ranges from 1 to 5 with higher scores reflecting greater gender awareness.
Time Frame: 24-month change in gender awareness among VA primary care and women's health providers and staff
Population: Primary care and women's health providers and staff. The analysis was based on cases with non-missing outcome data. There are 22 missing cases in the EBQI arm and 32 in the control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 246 | 439
Number analyzed (VA Medical Centers) | 7 | 14
score on a scale
  Baseline: number analyzed (Participants) | 124 | 217
  Baseline | 3.66 (0.53) | 3.63 (0.49)
  24-month: number analyzed (Participants) | 122 | 222
  24-month | 3.64 (0.51) | 3.74 (0.54)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Change in gender awareness score between EBQI and control from baseline to 24-month; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.29, Regression, Linear — P-value reflects the interaction term between EBQI and time, adjusted for non-response weights and characteristics described in the statistical analysis overview; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.33 to 0.10], Standard Error of Mean 0.10 — The estimated value reported here is the predicted mean change from baseline to 24-month, adjusting for characteristics described in the statistical analysis overview

5. Primary Outcome: Quality Improvement Experience
Description: The count of quality improvement activities reported by providers and staff in primary care and women's health settings; including 1) training in quality improvement methods, 2) collaboration with other VA facilities to identify best practices, 3) working with Women Veteran Program Manager to identify and/or solve local problems in caring for women Veterans, 4) using of VA performance data, 5) using of VA survey data by gender, 6) working on a quality improvement project focused on women Veterans, 7) involving in small tests of change for quality improvement.
Time Frame: 12-month change
Population: Primary care and women's health providers and staff at 21 VA Medical Centers. The analysis was based on cases with non-missing outcome data. There were 31 missing in the EBQI arm and 43 missing in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 205 | 422
Participants
  Baseline: number analyzed (Participants) | 124 | 217
  Baseline: 0 activity | 29 | 70
  Baseline: 1 activity | 17 | 46
  Baseline: 2 activities | 17 | 29
  Baseline: 3 activities | 11 | 19
  Baseline: 4 activities | 14 | 13
  Baseline: 5 activities | 3 | 4
  Baseline: 6 activities | 8 | 7
  Baseline: 7 activities | 2 | 4
  Baseline: missing | 23 | 25
  12-month: number analyzed (Participants) | 81 | 205
  12-month: 0 activity | 26 | 54
  12-month: 1 activity | 16 | 41
  12-month: 2 activities | 13 | 38
  12-month: 3 activities | 5 | 22
  12-month: 4 activities | 6 | 11
  12-month: 5 activities | 2 | 12
  12-month: 6 activities | 2 | 5
  12-month: 7 activities | 3 | 4
  12-month: missing | 8 | 18
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Superiority — Difference-in-differences analysis using logistic regression. The number of activities were recoded into 0 vs 1+ activities. The model was adjusted for age, how often they saw women patients in the past year, location of practice in primary care or women's health clinic, and having had any type of quality improvement training. We also adjusted for non-response weights; p = 0.10, Difference-in-Differences analysis — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = -0.69, 95% CI 2-sided [-1.52 to 0.13], Standard Error of Mean 0.42 — The estimated value is predicted change in the odds of involving in one or more quality improvement activities, adjusting for characteristics described in the statistical analysis overview

6. Primary Outcome: Quality Improvement Experience
Description: The count of quality improvement activities reported by provider and staff in primary care and women's health settings; including 1) training in quality improvement methods [e.g., LEAN], 2) collaboration with other VA facilities to identify best practices, 3) working with Women Veteran Program Manager to identify and/or solve local problems in caring for women Veterans, 4) using of VA performance data, 5) using of VA survey data by gender, 6) working on a quality improvement project focused on women Veterans, 7) involving in small tests of change for quality improvement.
Time Frame: 24-month change
Population: Primary care and women's health providers and staff at 21 VA Medical Centers. The analysis was based on cases with non-missing outcome data. There were 27 missing in the EBQI arm and 32 missing in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 246 | 439
Participants
  Baseline: number analyzed (Participants) | 124 | 217
  Baseline: 0 activity | 29 | 70
  Baseline: 1 activity | 17 | 46
  Baseline: 2 activities | 17 | 29
  Baseline: 3 activities | 11 | 19
  Baseline: 4 activities | 14 | 13
  Baseline: 5 activities | 3 | 4
  Baseline: 6 activities | 8 | 7
  Baseline: 7 activities | 2 | 4
  Baseline: missing | 23 | 25
  24-month: number analyzed (Participants) | 122 | 222
  24-month: 0 activity | 44 | 66
  24-month: 1 activity | 19 | 43
  24-month: 2 activities | 22 | 39
  24-month: 3 activities | 18 | 27
  24-month: 4 activities | 7 | 16
  24-month: 5 activities | 2 | 9
  24-month: 6 activities | 3 | 12
  24-month: 7 activities | 3 | 3
  24-month: missing | 4 | 7
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.22, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = -0.48, 95% CI 2-sided [-1.25 to 0.29], Standard Error of Mean 0.39 — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Gender-specific Preventive Care Delivery
Description: Rate of cervical cancer screening using the VA External Peer Review Program (EPRP) chart-based quality metrics.
Time Frame: 12-month change
Population: The analysis population size was extracted from EPRP reported denominators. EPRP randomly selected women patients aged 21-64and reviewed their charts for cervical cancer screening with a Pap test in the past three years.
Measure: Mean (Standard Deviation); unit: percentage of women patients
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 4077 | 7057
Number analyzed (VA Medical Centers) | 7 | 14
percentage of women patients
  Baseline: number analyzed (Participants) | 1975 | 3666
  Baseline | 87.5 (4.1) | 87.2 (4.3)
  12 month: number analyzed (Participants) | 2102 | 3391
  12 month | 87.5 (3.9) | 88.1 (6.11)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — Analysis of Variance testing the differences in outcome between EBQI and control groups over 12 month period; p = 0.788, ANOVA — The p-value reflects the interaction term between EBQI and time; Mean Difference (Net) = -0.08, 95% CI 2-sided [-7.1 to 5.4], Standard Error of Mean 3.1

8. Secondary Outcome: Gender-specific Preventive Care Delivery
Description: Rate of cervical cancer screening using the VA External Peer Review Program (EPRP) chart-based quality metrics.
Time Frame: 24-month change in gender-specific preventive care delivery
Population: The analysis population size is extracted from EPRP reported denominators. EPRP randomly selected women patients aged 21-64and reviewed their charts for cervical cancer screening with a Pap test in the past three years.
Measure: Mean (Standard Deviation); unit: percentage of women patients
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 3549 | 7733
Number analyzed (VA Medical Centers) | 7 | 14
percentage of women patients
  Baseline: number analyzed (Participants) | 1975 | 3666
  Baseline | 87.5 (4.12) | 87.2 (4.30)
  24 month: number analyzed (Participants) | 1574 | 4067
  24 month | 84.6 (3.98) | 85.8 (4.83)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — Analysis of Variance testing for differences in outcomes between EBQI and control arms from baseline to 24 months; p = 0.61, ANOVA — The p-value reflects the interaction terms between EBQI and control arms; Mean Difference (Net) = -1.5, 95% CI 2-sided [-7.35 to 4.35], Standard Error of Mean 2.89

9. Secondary Outcome: Accessibility of Care
Description: Women Veterans' ratings of accessibility based on the Survey of Healthcare Experience of Patients (SHEP) program. The mean score is the percent of female patients who responded "always" to validated survey items measuring accessibility, the higher percentage representing better access.
Time Frame: 12-month change in accessibility
Population: The analysis population size is extracted from SHEP, which randomly selected eligible patients who were invited to respond to the SHEP surveys by mail or online.
Measure: Mean (Standard Deviation); unit: percent always
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 315 | 495
Number analyzed (VA Medical Centers) | 7 | 14
percent always
  baseline: number analyzed (Participants) | 262 | 309
  baseline | 48.6 (12.2) | 44.4 (18.5)
  12month: number analyzed (Participants) | 53 | 186
  12month | 41.1 (24.5) | 37.1 (8.0)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — ANOVA comparing changes in outcome over time between EBQI and control arms; p = 0.987, ANOVA — The p-value reflects the interaction term between EBQI and time; Mean Difference (Net) = -0.17, 95% CI 2-sided [-21.45 to 21.11], Standard Error of Mean 10.5

10. Secondary Outcome: Accessibility of Care
Description: Women Veterans' ratings of accessibility from the Survey of Healthcare Experience of Patients (SHEP) program. The mean score is the percent of female patients who responded "always" to validated survey items measuring accessibility, the higher percentage representing better access.
Time Frame: 24-month change in accessibility
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percent always
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 340 | 466
Number analyzed (VA Medical Centers) | 7 | 14
Percent always
  Baseline: number analyzed (Participants) | 262 | 309
  Baseline | 46.7 (9.3) | 43.0 (17.8)
  24month: number analyzed (Participants) | 78 | 157
  24month | 42.7 (13.7) | 42.3 (14.7)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — ANOVA comparing changes in outcome over time between EBQI and control groups; p = 0.708, ANOVA — The p-value reflects the interaction terms between EBQI and time; Mean Difference (Net) = -3.91, 95% CI 2-sided [-24.89 to 17.08], Standard Error of Mean 10.35

11. Secondary Outcome: Coordination of Care
Description: Women Veterans' ratings of care coordination from the Survey of Healthcare Experience of Patients (SHEP) program. The mean score is the percent of female patients who responded "always" to validated survey items measuring care coordination, the higher percentage representing better coordination.
Time Frame: 12-month change
Population: The analysis population size is unknown and reported at the level of the VA Medical Centers. SHEP randomly selected eligible patients who were invited to respond to the SHEP surveys by mail or online.
Measure: Mean (Standard Deviation); unit: percent always
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 510 | 790
Number analyzed (VA Medical Centers) | 7 | 14
percent always
  baseline: number analyzed (Participants) | 422 | 486
  baseline | 54.60 (12.43) | 55.78 (14.05)
  12 month: number analyzed (Participants) | 88 | 304
  12 month | 52.95 (19.30) | 58.65 (9.67)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — ANOVA comparing changes in outcome over time between EBQI and control groups; p = 0.613, ANOVA — The p-value reflects the interaction term between EBQI and time; Mean Difference (Net) = -4.51, 95% CI 2-sided [-22.43 to 13.40], Standard Error of Mean 8.85

12. Secondary Outcome: Coordination of Care
Description: as for outcome 11
Time Frame: 24-month change
Population: The analysis population size is extracted SHEP, which randomly selected eligible patients who were invited to respond to the SHEP surveys by mail or online.
Measure: Mean (Standard Deviation); unit: percent always
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 541 | 750
Number analyzed (VA Medical Centers) | 7 | 14
percent always
  baseline: number analyzed (Participants) | 422 | 486
  baseline | 53.0 (9.3) | 54.7 (13.4)
  24 month: number analyzed (Participants) | 119 | 264
  24 month | 51.4 (13.7) | 51.2 (15.2)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — ANOVA comparing changes in outcome over time between EBQI and control groups; p = 0.922, ANOVA — The p-value reflects the interaction term between EBQI and time; Mean Difference (Net) = 0.94, 95% CI 2-sided [-18.26 to 20.13], Standard Error of Mean 9.48

13. Secondary Outcome: Gender-neutral Guideline-concordant Preventive Care Receipt
Description: Percentage of women Veterans' obtaining recommended preventive care based on eligibility for service (e.g., meet eligibility guidelines for timely eye exams for diabetes, flu vaccination, colorectal cancer screening) using VA External Peer Review Program (EPRP) chart-based quality metrics.
Time Frame: 12-month change
Population: The analysis population is extracted from EPRP, which randomly selected VA women patients aged 18-75 whose charts were reviewed for preventive care measures.
Measure: Mean (Standard Deviation); unit: percentage of female patients
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 43587 | 73735
Number analyzed (VA Medical Centers) | 7 | 14
percentage of female patients
  Baseline: number analyzed (Participants) | 21684 | 31334
  Baseline | 78.8 (2.2) | 78.6 (2.9)
  12 month: number analyzed (Participants) | 21907 | 42401
  12 month | 75.9 (4.7) | 75.1 (3.1)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — two-way ANOVA testing change in a composite score of gender-neutral preventive care between EBQI and control arms over time; p = 0.789, ANOVA — The p-value represents the interaction term between EBQI and control; Mean Difference (Net) = 0.58, 95% CI 2-sided [-3.74 to 4.89], Standard Error of Mean 2.13

14. Secondary Outcome: Gender-neutral Guideline-concordant Preventive Care Receipt
Description: as for outcome 13
Time Frame: 24-month change
Population: The analysis population is extracted from EPRP, which randomly selected women patients aged 18-75 whose charts were reviewed for preventive care metrics.
Measure: Mean (Standard Deviation); unit: percentage of female patients
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 39271 | 73819
Number analyzed (VA Medical Centers) | 7 | 14
percentage of female patients
  Baseline: number analyzed (Participants) | 21684 | 31334
  Baseline | 78.8 (2.23) | 78.6 (2.75)
  24 month: number analyzed (Participants) | 17587 | 45485
  24 month | 75.9 (4.7) | 75.0 (3.0)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — ANOVA comparing changes in outcomes over time between EBQI and control groups; p = 0.51, ANOVA — The p-value reflects the interaction between EBQI and time; The analysis is adjusted for EBQI and time; Mean Difference (Net) = -1.63, 95% CI 2-sided [-6.60 to 3.33], Standard Error of Mean 2.45

15. Secondary Outcome: Assignment to a Designated Women's Health Provider or a Women's Health Primary Care Teams, Using Patient Aligned Care Teams Compass
Description: Percentage of women Veterans assigned to a designated women's health provider in a general primary care and/or women's health primary care setting.
Time Frame: 12-month change
Population: The analysis population was extracted from the Patient Aligned Care Teams (PACT) Compass, developed to meet the needs for VA PACT implementation.
Measure: Mean (Standard Deviation); unit: percentage of female patients
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 82328 | 127153
Number analyzed (VA Medical Centers) | 7 | 14
percentage of female patients
  Baseline: number analyzed (Participants) | 39664 | 61513
  Baseline | 65.8 (17.2) | 65.8 (17.2)
  12 month: number analyzed (Participants) | 42664 | 65640
  12 month | 74.0 (6.3) | 73.8 (13.7)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — ANOVA testing for change in outcome over time between EBQI and control arms; p = 0.711, ANOVA — The p-value reflects the interaction between EBQI and time; Mean Difference (Net) = 3.11, 95% CI 2-sided [-13.7 to 19.9], Standard Error of Mean 8.3

16. Secondary Outcome: Assignment to a Designated Women's Health Provider or a Women's Health Primary Care Teams, Using Patient Aligned Care Teams Compass
Description: as for outcome 15
Time Frame: 24-month change
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage of female patients
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 64461 | 151493
Number analyzed (VA Medical Centers) | 7 | 14
percentage of female patients
  Baseline: number analyzed (Participants) | 39664 | 61513
  Baseline | 65.8 (17.2) | 68.7 (11.3)
  24 month: number analyzed (Participants) | 24797 | 89980
  24 month | 78.6 (11.3) | 73.1 (13.8)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — ANOVA comparing changes in outcome over time between EBQI and control arms; p = 0.335, ANOVA — The p-value reflects the interaction term between EBQI and time; Mean Difference (Net) = 8.49, 95% CI 2-sided [-9.1 to 26.1], Standard Error of Mean 8.7

17. Secondary Outcome: Provider Rating
Description: Percent of women patients who rated 9 or 10 on a scale of 0 to 10 for the provider rating question on the Survey of Healthcare Experiences of Patients (SHEP). Higher scores are better.
Time Frame: 12 month change
Population: Analysis population size was extracted SHEP, which randomly selected eligible patients who were invited to respond to the SHEP surveys by mail or online.
Measure: Mean (Standard Deviation); unit: percentage of women patients
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 535 | 832
Number analyzed (VA Medical Centers) | 7 | 14
percentage of women patients
  Baseline: number analyzed (Participants) | 443 | 513
  Baseline | 65.9 (13.5) | 63.6 (16.7)
  12 Month: number analyzed (Participants) | 92 | 319
  12 Month | 59.9 (32.5) | 71.3 (13.4)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — Analysis of Variance testing for change in outcome between EBQI and control groups from baseline to 12 months; p = 0.268, ANOVA — P-value is from the interaction term between EBQI and time; Mean Difference (Net) = -13.8, 95% CI 2-sided [-38.7 to 11.1], Standard Error of Mean 12.3

18. Secondary Outcome: Provider Rating
Description: Percent of women patients who rated 9 or 10 on a scale of 0 to 10 for the provider rating question from the Survey of Healthcare Experiences of Patients (SHEP). Higher scores are better.
Time Frame: 24-month change
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of women patients
Units Other Than Participants: VA Medical Centers
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
Number analyzed (Participants) | 571 | 786
Number analyzed (VA Medical Centers) | 7 | 14
percentage of women patients
  Baseline: number analyzed (Participants) | 443 | 513
  Baseline | 65.9 (13.5) | 63.6 (16.7)
  24 months: number analyzed (Participants) | 128 | 273
  24 months | 59.7 (14.2) | 57.5 (14.2)
Statistical Analysis 1: Comparison: Evidence-Based Quality Improvement (EBQI) vs Waitlist Controls; Test type: Non-Inferiority — Analysis of Variance testing the differences between EBQI and control from baseline and 24 months; p = 0.991, ANOVA — P-value is from the interaction between EBQI and time; Mean Difference (Net) = -0.14, 95% CI 2-sided [-25.6 to 25.3], Standard Error of Mean 12.6

ADVERSE EVENTS:
Time Frame: Study time frame was over three years (fiscal years 2017, 2018, 2019).
Description: Adverse events (all-cause mortality, serious adverse events, other adverse events) were not monitored/assessed for this study as the target of EBQI was the VA facility and the providers and staff therein. Data collection focused on surveys about their attitudes (e.g., gender sensitivity) and experiences with and perspectives on quality improvement for comprehensive women's health care.
Arm/Group | Evidence-Based Quality Improvement (EBQI) | Waitlist Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT03238417/Prot_SAP_000.pdf